CLINICAL TRIAL: NCT00210652
Title: A Double-Blind, Placebo-Controlled, Dose-Titration Study to Determine Safety, Tolerability and Preliminary Efficacy of RWJ-333369 as Adjunctive Therapy in Subjects With Treatment-Resistant Partial Seizures (With or Without Secondary Generalization) or Primarily Generalized Tonic-Clonic Seizures
Brief Title: An Open-Label Extension Study to Evaluate the Safety and Effectiveness of RWJ 333369 in Patients With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004147
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Epilepsy; Epilepsies, Partial
Keywords: Epilepsy; Refractory partial epilepsy; seizure disorder; antiepileptic drugs
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

ARMS (1):
- 001 (Experimental): RWJ 333369: Open-Label Extension: One 250mg tablet twice daily up to a total of 1200mg/day up until RWJ-33369 is available by prescription or study is terminated by sponsor
  Interventions: Drug: RWJ 333369:

INTERVENTIONS:
Drug: RWJ 333369: — Open-Label Extension: One 250mg tablet twice daily up to a total of 1200mg/day up until RWJ-33369 is available by prescription or study is terminated by sponsor

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary effectiveness of the novel compound RWJ-333369 in patients with partial onset seizures who are currently being treated with 1 or 2 concomitant antiepileptic drugs.

DETAILED DESCRIPTION:
333369EPY2002 is the open-label extension study that follows the double-blind study 333369EPY2001. In an open label study such as 333369EPY2002, both the physician and the patient know the name of the assigned study medication. In a double blind study such as 333369EPY2001, neither the physician nor the patient knows the name of the assigned study medication. Patients who complete the double-blind treatment phase of study 333369EPY2001 will be eligible to enter the open-label extension study during which patients will transition through a blinded period to an open-label period with carisbamate (also referred to as RWJ-333369). RWJ-333369 is a new chemical compound with anticonvulsant activity that is currently under investigation as a treatment for epilepsy. Patients electing to enter the open-label extension phase will be supplied with both open-label carisbamate (RWJ-333369) and blinded study medication for the transition phase. During this transition phase (up to 21 days in length), the patient's dose of double-blind study drug will be gradually reduced and stopped and treatment with open-label RWJ-333369 will be started. Throughout the remainder of the open label extension phase, investigators will be allowed to make further adjustments of the dosage and schedule of carisbamate, including independent adjustment of the morning and evening doses, but a dosage of 1,200 mg/day may not be exceeded and increases in dosage must be in increments of no more than 200 mg/day. Patients who, in the judgment of the investigator, continue to benefit from treatment with RWJ-333369 may continue to receive the drug with follow up clinic visits every 3 months until RWJ 333369 is available by prescription or the program is terminated by the sponsor. Initial dose RWJ-333369 is 1 capsule (250 milligram (mg) taken twice daily. Dosage may be changed at weekly intervals. The maximum permitted dose will be 4 capsules (1000 mg), twice daily during dose titration. Double blind-treatment duration is up to 71 days with the option to continue treatment in an open-label study. Maximum dose in open-label study is 1200 mg/day

ELIGIBILITY:
Inclusion Criteria:

* In order to enter the open label extension, the patient must have completed Study 333369EPY-2001.

Exclusion Criteria:

* Patients who have seizures that cannot be quantitated accurately
* patients with a history of nonepileptic seizures, serious systemic disease, progressive neurologic disorder, a major psychiatric disorder, status epilepticus in the past 3 months, vagal nerve stimulation discontinuation within the past 3 months
* patients with a history of drug or alcohol abuse within the past 2 years
* patients currently taking felbamate, vigabatrin, or tricyclic antidepressants
* and female patients who are pregnant or nursing.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Adverse events as a measure of safety and tolerability | At followup visits every 3 months up to the time RWJ-333369 is available by prescription or study is terminated by sponsor

SECONDARY OUTCOMES:
Seizure counts | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.